CLINICAL TRIAL: NCT01559935
Title: A Phase II Study of Sequential Carfilzomib, Clarithromycin (Biaxin®), Lenalidomide (Revlimid®), and Dexamethasone (Decadron®) [Car-BiRD] Therapy for Subjects With Newly Diagnosed Multiple Myeloma
Brief Title: Carfilzomib, Clarithromycin (Biaxin®), Lenalidomide (Revlimid®), and Dexamethasone (Decadron®) [Car-BiRD] Therapy for Subjects With Multiple Myeloma
Acronym: CarBiRD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1108011903
Record Dates: First submitted 2012-02-16; First posted 2012-03-21 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; Clarithromycin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Car-BiRD Therapy (Experimental): Carfilzomib, Clarithromycin (Biaxin®), Lenalidomide (Revlimid®), and Dexamethasone (Decadron®) [Car-BiRD]
  Interventions: Drug: carfilzomib; Drug: Dexamethasone; Drug: Clarithromycin; Drug: Lenalidomide

INTERVENTIONS:
Drug: carfilzomib — 45 mg/m2 IV on days 1, 2, 8, 9, 15 and 16 of each 28 day cycles.
Drug: Dexamethasone — 20 mg orally on days 1, 2, 8, 9, 15 and 16 of a 28 day cycle, while receiving carfilzomib.
  Other Names: DECADRON®
Drug: Clarithromycin — 500 mg twice a day for each 28 day cycle of BiRD treatment. BiRD begins after carfilzomib treatment has been completed.
  Other Names: Biaxin
Drug: Lenalidomide — 25 mg orally days 1-21 for each 28 day cycle of BiRD treatment. BiRD begins after carfilzomib treatment has been completed.
  Other Names: Revlimid
Drug: Dexamethasone — 40 mg orally on days 1, 8, 15 and 22 of each 28 day cycle of BiRD treatment. BiRD begins after carfilzomib treatment has been completed.
Drug: Lenalidomide — 10 mg orally on days 1-21 or each 28 day cycle of maintenance. Maintenance begins after BiRD treatment has been completed.
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an investigational new drug called carfilzomib, in combination with dexamethasone in subjects with newly diagnosed multiple myeloma followed by treatment with a combination of drugs clarithromycin (Biaxin®), lenalidomide (Revlimid®) and dexamethasone (Decadron®) [BiRD] then lenalidomide alone.

DETAILED DESCRIPTION:
While new anti-myeloma therapies such as bortezomib and immunomodulatory drugs have been developed, multiple myeloma remains an incurable malignancy. Given that obtaining a complete remission (CR) with therapy will allow patients with newly diagnosed multiple myeloma to enjoy a higher quality of life and longer duration of freedom from disease symptoms, finding an optimally effective and well-tolerated regimen is imperative.

The robust overall response rate of 91% with the BiRD regimen for patients with newly diagnosed multiple myeloma is encouraging and we believe that by adding carfilzomib the overall response rate and CR rate can be improved. As carfilzomib has proven efficacy in myeloma and in patient's who have relapsed on bortezomib, we anticipate that it will synergize with the previous BiRD regimen to induce greater reduction of tumor burden overall.

The primary endpoints include best response rate, toxicities, progression free survival, event free survival, and overall survival. In those patients who are eligible for autologous stem cell transplantation, we will also study the effect of carfilzomib on CD 34+ stem cell yield following mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Subject is ≥ 18 years at the time of signing the consent form.
* Subject has histologically confirmed multiple myeloma that has never before been treated.
* Subject had no anti-myeloma therapy within 14 days prior to initiation of study treatment except for corticosteroids with a maximum allowed dosage equivalent to three pulses of dexamethasone (40mg daily for 4 days equals one pulse). Patients may have received prior adjuvant antiresorptive therapy (i.e., pamidronate or zoledronic acid) as routine care, or radiation therapy as palliation for pain and/or spinal cord compression.
* Subject has measurable disease as defined by > 0.5 g/dL serum monoclonal protein, > 10 mg/dL involved serum free light chain (either kappa or lambda) provided that the serum free light chain ratio is abnormal, > 0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s) of at least 1cm in greatest dimension as measured by either CT scanning or MRI.
* Subject has a Karnofsky performance status ≥ 60% (> 50% if due to bony involvement of myeloma (see Appendix VI).
* Subject is able to take prophylactic anticoagulation as detailed in section 9.1 (patients intolerant to aspirin may use warfarin or low molecular weight heparin).
* Subject is registered into the mandatory RevAssist® program, and is willing and able to comply with the requirements of RevAssist® program.
* If subject is a female of childbearing potential (FCBP),† she must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy.
* Subjects must meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L)
  * Hemoglobin ≥ 7 g/dL
  * Platelet count ≥ 30,000/mm3 (75 x 109/L)
  * Serum SGOT/AST < 3.0 x upper limits of normal (ULN)
  * Serum SGPT/ALT < 3.0 x upper limits of normal (ULN)
  * Serum creatinine < 2.5 mg/dL (221 µmol/L)
  * Serum total bilirubin < 2.0 mg/dL (34 µmol/L)

Exclusion Criteria:

* Subject has immeasurable MM (no measurable monoclonal protein, free light chains in blood or urine, or measureable plasmacytoma on radiologic scanning).
* Subject has a prior history of other malignancies unless disease free for ≥ 5 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or localized prostate cancer with Gleason score < 7 with stable prostate specific antigen (PSA) levels.
* Subject has had myocardial infarction within 6 months prior to enrollment , or NYHA(New York Hospital Association) Class III or IV heart failure, Ejection Fraction < 35%, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Female subject who is pregnant or lactating.
* Subject has known HIV infection
* Subject has known active hepatitis B or hepatitis C infection.
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Subject has known hypersensitivity to dexamethasone, clarithromycin, lenalidomide, thalidomide, allopurinol, or carfilzomib.
* Subject has a history of thromboembolic event within the past 4 weeks prior to enrollment.
* Subject has any clinically significant medical or psychiatric disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-04-19 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2027-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were ineligible and therefore never started treatment.
Groups:
- Car-BiRD Therapy: Carfilzomib, Clarithromycin (Biaxin®), Lenalidomide (Revlimid®), and Dexamethasone (Decadron®) [Car-BiRD]
  Car Phase:
  carfilzomib: 45 mg/m2 IV on days 1, 2, 8, 9, 15 and 16 of each 28 day cycles. Dexamethasone: 20 mg orally on days 1, 2, 8, 9, 15 and 16 of a 28 day cycle, while receiving carfilzomib.
  BiRD Phase:
  Clarithromycin: 500 mg twice a day for each 28 day cycle of BiRD treatment. BiRD begins after carfilzomib treatment has been completed.
  Lenalidomide: 25 mg orally days 1-21 for each 28 day cycle of BiRD treatment. BiRD begins after carfilzomib treatment has been completed.
  Dexamethasone: 40 mg orally on days 1, 8, 15 and 22 of each 28 day cycle of BiRD treatment. BiRD begins after carfilzomib treatment has been completed.
  Maintenance Phase:
  Lenalidomide: 10 mg orally on days 1-21 or each 28 day cycle of maintenance. Maintenance begins after BiRD treatment has been completed.
Period: Car Phase
Arm/Group | Car-BiRD Therapy
Started | 72
Completed | 58
Not Completed | 14
Not completed — Toxicity | 4
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Per protocol | 1
Not completed — Insurance | 1
Not completed — non-compliance | 1
Period: BiRD Phase
Arm/Group | Car-BiRD Therapy
Started | 58
Completed | 54
Not Completed | 4
Not completed — Toxicity | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 2
Period: Maintenance Phase
Arm/Group | Car-BiRD Therapy
Started | 54
Completed | 0
Not Completed | 54
Not completed — Remains on study | 28
Not completed — Toxicity | 1
Not completed — Lack of Efficacy | 18
Not completed — Withdrawal by Subject | 5
Not completed — Non-compliance | 2

BASELINE CHARACTERISTICS:
Population: 72 subjects started the Car Phase of the CarBiRD therapy. 58 subjects started the BiRD Phase of the CarBiRD therapy. 54 subjects started the Maintenance Phase of the CarBiRD therapy. A detailed explanation of those numbers is provided in the participant flow.
Arm/Group | Car-BiRD Therapy
Number analyzed (Participants) | 72
Age, Customized [Mean (Full Range); unit: years] — Population: 72 subjects started the Car Phase of the CarBiRD therapy. 58 subjects reached the BiRD Phase of the CarBiRD therapy. 54 subjects reached the Maintenance Phase of the CarBiRD therapy. A detailed explanation of those numbers is provided in the participant flow.
  years
    Car Phase | 60.4 [42 to 85]
    BiRD Phase: number analyzed (Participants) | 58
    BiRD Phase | 59.6 [42 to 85]
    Maintenance Phase: number analyzed (Participants) | 54
    Maintenance Phase | 59.2 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 72 subjects started the Car Phase of the CarBiRD therapy. 58 subjects reached the BiRD Phase of the CarBiRD therapy. 54 subjects reached the Maintenance Phase of the CarBiRD therapy. A detailed explanation of those numbers is provided in the participant flow.
  Participants
    Car Phase: Female | 29
    Car Phase: Male | 43
    BiRD Phase: number analyzed (Participants) | 58
    BiRD Phase: Female | 26
    BiRD Phase: Male | 32
    Maintenance Phase: number analyzed (Participants) | 54
    Maintenance Phase: Female | 23
    Maintenance Phase: Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 72 subjects started the Car Phase of the CarBiRD therapy. 58 subjects started the BiRD Phase of the CarBiRD therapy. 54 subjects started the Maintenance Phase of the CarBiRD therapy. A detailed explanation of those numbers is provided in the participant flow.
  Participants
    Car Phase: Hispanic or Latino | 3
    Car Phase: Not Hispanic or Latino | 61
    Car Phase: Unknown or Not Reported | 8
    BiRD Phase: number analyzed (Participants) | 58
    BiRD Phase: Hispanic or Latino | 3
    BiRD Phase: Not Hispanic or Latino | 48
    BiRD Phase: Unknown or Not Reported | 7
    Maintenance Phase: number analyzed (Participants) | 54
    Maintenance Phase: Hispanic or Latino | 2
    Maintenance Phase: Not Hispanic or Latino | 45
    Maintenance Phase: Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 72 subjects started the Car Phase of the CarBiRD therapy. 58 subjects started the BiRD Phase of the CarBiRD therapy. 54 subjects started the Maintenance Phase of the CarBiRD therapy. A detailed explanation of those numbers is provided in the participant flow.
  Participants
    Car Phase: American Indian or Alaska Native | 0
    Car Phase: Asian | 0
    Car Phase: Native Hawaiian or Other Pacific Islander | 0
    Car Phase: Black or African American | 5
    Car Phase: White | 29
    Car Phase: More than one race | 6
    Car Phase: Unknown or Not Reported | 32
    BiRD Phase: number analyzed (Participants) | 58
    BiRD Phase: American Indian or Alaska Native | 0
    BiRD Phase: Asian | 0
    BiRD Phase: Native Hawaiian or Other Pacific Islander | 0
    BiRD Phase: Black or African American | 4
    BiRD Phase: White | 22
    BiRD Phase: More than one race | 5
    BiRD Phase: Unknown or Not Reported | 27
    Maintenance Phase: number analyzed (Participants) | 54
    Maintenance Phase: American Indian or Alaska Native | 0
    Maintenance Phase: Asian | 0
    Maintenance Phase: Native Hawaiian or Other Pacific Islander | 0
    Maintenance Phase: Black or African American | 3
    Maintenance Phase: White | 20
    Maintenance Phase: More than one race | 5
    Maintenance Phase: Unknown or Not Reported | 26

OUTCOME MEASURES:

1. Primary Outcome: Response to Car-BiRD Treatment.
Description: The best response for all patients who had at least one dose of drug was measured.
  Response categories:
  Stringent Complete Response (sCR), Complete Remission(CR), Very Good Partial Remission(VGPR), Partial Remission (PR), Progressive Disease (PD), Stable Disease (SD).
  The response is evaluated based on the IMWG criteria.
Time Frame: From baseline to best response, up to 116 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Car-BiRD Therapy
Number analyzed (Participants) | 72
Participants
  sCR/CR | 28
  VGPR | 31
  PR | 11
  SD | 1
  PD | 0
  Not Evaluable | 1

2. Secondary Outcome: Event Free Survival
Description: an event is defined by coming off protocol for any reason, including progression of disease, lack of disease response, regimen intolerability, withdrawal of consent or death.
Time Frame: From date of study enrollment until the date of removal of study due to progression of disease, toxicity or withdrawal of consent, up to 1222 days.
Population: 44 participants analyzed out of the 72 participants initially enrolled in the study. 28 participants are active and therefore have not experienced any events leading to removal from study.
Measure: Median (Full Range); unit: Days
Arm/Group | Car-BiRD Therapy
Number analyzed (Participants) | 44
Days | 401.5 [18 to 1222]

3. Secondary Outcome: MRD Negativity Following CarBiRD Regimen
Description: Minimal Residual Disease (MRD) was assessed for all participants as soon as they achieved CR/sCR, regardless of what phase they were on.
  MRD negativity is defined as the complete absence of plasma cells on bone marrow biopsy.
  MRD positivity is defined as the presence of residual plasma cells (<5%) on bone marrow biopsy.
  The IMWG criteria were used to determine CR and sCR.
Time Frame: From start of study up to Revlimid Maintenance Cycle 4.
Population: 28 participants achieved CR or sCR.
Measure: Count of Participants; unit: Participants
Arm/Group | Car-BiRD Therapy
Number analyzed (Participants) | 28
Participants
  MRD positive | 10
  MRD negative | 17
  Not Evaluable | 1

4. Secondary Outcome: Progression Free Survival
Description: Progression was defined using the IMWG criteria.
Time Frame: From start of study drug until first incidence of progression, up to 1222 days.
Population: 21 participants had an incidence of progression.
Measure: Median (Full Range); unit: months
Arm/Group | Car-BiRD Therapy
Number analyzed (Participants) | 21
months | 18.3 [2.3 to 40.7]

5. Secondary Outcome: Stem Cells Collection
Description: At the end of the Car Phase, all participants underwent stem cell collection.
Time Frame: At the end of the Car Phase, prior to the start of the BiRD Phase, on average after 162 days.
Population: 58 participants reached the end of the Car Phase. From those 58 participants, 52 were collected, 5 participants declined stem cell collection and 1 participant's results were not evaluable.
Measure: Mean (Standard Deviation); unit: Number of stem cells collected per Kg
Arm/Group | Car-BiRD Therapy
Number analyzed (Participants) | 52
Number of stem cells collected per Kg | 12854635 (5388946.9)

ADVERSE EVENTS:
Description: Collection of adverse events is ongoing as 28 participants are still on trial.
  For the Car Phase, every adverse event not present at baseline was reported. For the BiRD and Maintenance phases, adverse events were only reported if it was a new occurrence (not present in the previous phase) or if the grade of the event increased.
  Grading was done using the CTCAE 4.0.
Arm/Group | Car-BiRD Therapy
All-Cause Mortality (participants affected / at risk) | 1/72
Serious Adverse Events (participants affected / at risk) | 26/72
Other Adverse Events (participants affected / at risk) | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Car-BiRD Therapy (N=72)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — car phase
fever (Vascular disorders) | 2 (3) — car phase
abnominal infection (Infections and infestations) | 1 (2) — car phase
lung infection (Infections and infestations) | 3 (4) — car phase
URI (Infections and infestations) | 2 (2) — car phase
UTI (Infections and infestations) | 2 (2) — car phase
femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — car phase
spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — car phase
atrial fibrilation (Cardiac disorders) | 1 (1) — car phase
massive heart attack (Cardiac disorders) | 1 (1) — car phase
syncope (Nervous system disorders) | 1 (1) — car phase
fall (Injury, poisoning and procedural complications) | 1 (1) — car phase
surgical procedure (Surgical and medical procedures) | 1 (1) — car phase
increased creatinine (Metabolism and nutrition disorders) | 1 (1) — car phase
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — car phase
dehydration (Metabolism and nutrition disorders) | 1 (1) — car phase
confusion (Nervous system disorders) | 1 (1) — car phase
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — car phase
thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — car phase
non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1/58 (1) — BiRD phase
abdominal pain (small intestinal obstruction) (Musculoskeletal and connective tissue disorders) | 1/58 (1) — BiRD phase
acute coronary syndrome (Cardiac disorders) | 1/58 (1) — BiRD phase
lung infection (Infections and infestations) | 3/58 (3) — BiRD phase
thromboembolic event (Vascular disorders) | 1/54 (1) — Maintenance phase
non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3/54 (3) — Maintenance phase
lung infection (Infections and infestations) | 4/54 (4) — Maintenance phase
diarrhea (Gastrointestinal disorders) | 1/54 (2) — Maintenance phase
acute kidney infection (Infections and infestations) | 1/54 (1) — Maintenance phase
enterocolitis infection (Infections and infestations) | 1/54 (1) — Maintenance phase
cardiac chest pain (Cardiac disorders) | 1/54 (1) — Maintenance phase
spinal cord compression (Musculoskeletal and connective tissue disorders) | 1/54 (1) — Maintenance phase
creatinine increase (Metabolism and nutrition disorders) | 1/54 (1) — Maintenance phase
secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/54 (1) — Maintenance phase
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Car-BiRD Therapy (N=72)
anemia (Blood and lymphatic system disorders) | 52 — Car phase
thrombocytopenia (Blood and lymphatic system disorders) | 64 — Car phase
neutropenia (Blood and lymphatic system disorders) | 13 — Car phase
leukopenia (Blood and lymphatic system disorders) | 25 — Car phase
lymphopenia (Blood and lymphatic system disorders) | 69 — Car phase
dyspepsia (Gastrointestinal disorders) | 13 — Car phase
constipation (Gastrointestinal disorders) | 18 — Car phase
nausea (Gastrointestinal disorders) | 17 — Car phase
anorexia (Gastrointestinal disorders) | 6 — Car phase
diarhhea (Gastrointestinal disorders) | 25 — Car phase
vomiting (Gastrointestinal disorders) | 8 — Car phase
flatulance (Gastrointestinal disorders) | 7 — Car phase
hypocalcemia (Metabolism and nutrition disorders) | 56 — Car phase
hyponatremia (Metabolism and nutrition disorders) | 42 — Car phase
hypoglycemia (Metabolism and nutrition disorders) | 21 — Car phase
hyperglycemia (Metabolism and nutrition disorders) | 63 — Car phase
hypophosphatemia (Metabolism and nutrition disorders) | 35 — Car phase
hyperkalemia (Metabolism and nutrition disorders) | 20 — Car phase
hypokalemia (Metabolism and nutrition disorders) | 4 — Car phase
hypomagnesemia (Metabolism and nutrition disorders) | 14 — Car phase
hypermagnesemia (Metabolism and nutrition disorders) | 10 — Car phase
hypoalbuminemia (Metabolism and nutrition disorders) | 39 — Car phase
hyperbilirubinemia (Metabolism and nutrition disorders) | 23 — Car phase
hyperuricemia (Metabolism and nutrition disorders) | 5 — Car phase
hyperhidrosis (Metabolism and nutrition disorders) | 8 — Car phase
elevated ALT (Metabolism and nutrition disorders) | 26 — Car phase
elevated AST (Metabolism and nutrition disorders) | 30 — Car phase
elevated alkaline phosphatase (Metabolism and nutrition disorders) | 34 — Car phase
increased creatinine (Metabolism and nutrition disorders) | 35 — Car phase
insomnia (General disorders) | 27 — Car phase
fatigue (General disorders) | 22 — Car phase
chills (General disorders) | 4 — Car phase
peripheral neuropathy (Nervous system disorders) | 12 — Car phase
tremor (Nervous system disorders) | 10 — Car phase
anxiety/stress (Nervous system disorders) | 13 — Car phase
depression (Psychiatric disorders) | 6 — Car phase
dizziness / lightheaded (Nervous system disorders) | 9 — Car phase
paresthesias (Nervous system disorders) | 4 — Car phase
forgetful (Nervous system disorders) | 4 — Car phase
dysgeusia (Nervous system disorders) | 4 — Car phase
headache (Nervous system disorders) | 12 — Car phase
irritability (Nervous system disorders) | 5 — Car phase
agitation (Nervous system disorders) | 4 — Car phase
concentration impairment (Nervous system disorders) | 7 — Car phase
edema (Vascular disorders) | 14 — Car phase
hypertension (Vascular disorders) | 4 — Car phase
fever (Vascular disorders) | 14 — Car phase
muscle spasms/cramps (Musculoskeletal and connective tissue disorders) | 13 — Car phase
muscle weakness (Musculoskeletal and connective tissue disorders) | 6 — Car phase
pain in legs (Musculoskeletal and connective tissue disorders) | 8 — Car phase
hip pain (Musculoskeletal and connective tissue disorders) | 7 — Car phase
back pain (Musculoskeletal and connective tissue disorders) | 17 — Car phase
knee pain (Musculoskeletal and connective tissue disorders) | 4 — Car phase
lower extremity pain (Musculoskeletal and connective tissue disorders) | 4 — Car phase
rash (Skin and subcutaneous tissue disorders) | 7 — Car phase
high BNP (Cardiac disorders) | 10 — Car phase
low eGFR (Renal and urinary disorders) | 37 — Car phase
genitourinary frequency (Renal and urinary disorders) | 4 — Car phase
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 — Car phase
cough (Respiratory, thoracic and mediastinal disorders) | 12 — Car phase
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 10 — Car phase
sore throat (Respiratory, thoracic and mediastinal disorders) | 4 — Car phase
URI (Infections and infestations) | 12 — Car phase
UTI (Infections and infestations) | 5 — Car phase
Skin Infection (Infections and infestations) | 4 — Car phase
neutropenia (Blood and lymphatic system disorders) | 6/58 — BiRD phase
leukopenia (Blood and lymphatic system disorders) | 5/58 — BiRD phase
lymphopenia (Blood and lymphatic system disorders) | 5/58 — BiRD phase
dyspepsia (Gastrointestinal disorders) | 4/58 — BiRD phase
constipation (Gastrointestinal disorders) | 15/58 — BiRD phase
nausea (Gastrointestinal disorders) | 7/58 — BiRD phase
anorexia (Gastrointestinal disorders) | 4/58 — BiRD phase
diarhhea (Gastrointestinal disorders) | 4/58 — BiRD phase
vomiting (Gastrointestinal disorders) | 3/58 — BiRD phase
dry mouth (Gastrointestinal disorders) | 4/58 — BiRD phase
flatulance (Gastrointestinal disorders) | 3/58 — BiRD phase
hypocalcemia (Metabolism and nutrition disorders) | 6/58 — BiRD phase
hypoglycemia (Metabolism and nutrition disorders) | 14/58 — BiRD phase
hypokalemia (Metabolism and nutrition disorders) | 4/58 — BiRD phase
hypomagnesemia (Metabolism and nutrition disorders) | 7/58 — BiRD phase
elevated ALT (Metabolism and nutrition disorders) | 3/58 — BiRD phase
ALK increase (Metabolism and nutrition disorders) | 6/58 — BiRD phase
increased creatinine (Metabolism and nutrition disorders) | 4/58 — BiRD phase
insomnia (General disorders) | 5/58 — BiRD phase
malaise (General disorders) | 3/58 — BiRD phase
fatigue (General disorders) | 9/58 — BiRD phase
peripheral neuropathy (Nervous system disorders) | 3/58 — BiRD phase
tremor (Nervous system disorders) | 11/58 — BiRD phase
dizziness / lightheaded (Nervous system disorders) | 5/58 — BiRD phase
parethesias (Nervous system disorders) | 4/58 — BiRD phase
dysgeusia (Nervous system disorders) | 17/58 — BiRD phase
irritability (Nervous system disorders) | 7/58 — BiRD phase
edema (Vascular disorders) | 10/58 — BiRD phase
cushingoid appearance (Vascular disorders) | 3/58 — BiRD phase
muscle spasms/cramps (Musculoskeletal and connective tissue disorders) | 6/58 — BiRD phase
hip pain (Musculoskeletal and connective tissue disorders) | 3/58 — BiRD phase
bone pain (Musculoskeletal and connective tissue disorders) | 3/58 — BiRD phase
rash (Skin and subcutaneous tissue disorders) | 13/58 — BiRD phase
pruritus (Skin and subcutaneous tissue disorders) | 3/58 — BiRD phase
low eGFR (Renal and urinary disorders) | 4/58 — BiRD phase
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3/58 — BiRD phase
lung infection (Respiratory, thoracic and mediastinal disorders) | 3/58 — BiRD phase
cough (Respiratory, thoracic and mediastinal disorders) | 3/58 — BiRD phase
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3/58 — BiRD phase
thrombocytopenia (Blood and lymphatic system disorders) | 3/54 — Maintenance phase
neutropenia (Blood and lymphatic system disorders) | 18/54 — Maintenance phase
leukopenia (Blood and lymphatic system disorders) | 11/54 — Maintenance phase
dyspepsia (Gastrointestinal disorders) | 13/54 — Maintenance phase
constipation (Gastrointestinal disorders) | 5/54 — Maintenance phase
nausea (Gastrointestinal disorders) | 4/54 — Maintenance phase
diarhhea (Gastrointestinal disorders) | 20/54 — Maintenance phase
vomiting (Gastrointestinal disorders) | 7/54 — Maintenance phase
dry mouth (Gastrointestinal disorders) | 3/54 — Maintenance phase
flatulance (Gastrointestinal disorders) | 3/54 — Maintenance phase
hypocalcemia (Metabolism and nutrition disorders) | 7/54 — Maintenance phase
hypercalcemia (Metabolism and nutrition disorders) | 3/54 — Maintenance phase
hypoglycemia (Metabolism and nutrition disorders) | 7/54 — Maintenance phase
hypophosphatemia (Metabolism and nutrition disorders) | 5/54 — Maintenance phase
hypokalemia (Metabolism and nutrition disorders) | 4/54 — Maintenance phase
hypomagnesemia (Metabolism and nutrition disorders) | 13/54 — Maintenance phase
hypoalbuminemia (Metabolism and nutrition disorders) | 8/54 — Maintenance phase
hyperbilirubinemia (Metabolism and nutrition disorders) | 5/54 — Maintenance phase
hyponatremia (Metabolism and nutrition disorders) | 3/54 — Maintenance phase
hypernatremia (Metabolism and nutrition disorders) | 5/54 — Maintenance phase
elevated ALT (Metabolism and nutrition disorders) | 5/54 — Maintenance phase
elevated AST (Metabolism and nutrition disorders) | 4/54 — Maintenance phase
increased creatinine (Metabolism and nutrition disorders) | 7/54 — Maintenance phase
fatigue (General disorders) | 5/54 — Maintenance phase
gait disturbance (General disorders) | 4/54 — Maintenance phase
hair loss (General disorders) | 4/54 — Maintenance phase
peripheral neuropathy (Nervous system disorders) | 7/54 — Maintenance phase
anxiety/stress (Psychiatric disorders) | 3/54 — Maintenance phase
depression (Psychiatric disorders) | 5/54 — Maintenance phase
dizziness / lightheaded (Nervous system disorders) | 5/54 — Maintenance phase
headache (Nervous system disorders) | 3/54 — Maintenance phase
edema (Vascular disorders) | 14/54 — Maintenance phase
hypertension (Vascular disorders) | 5/54 — Maintenance phase
muscle spasms/cramps (Musculoskeletal and connective tissue disorders) | 5/54 — Maintenance phase
shoulder pain (Musculoskeletal and connective tissue disorders) | 5/54 — Maintenance phase
rib pain (Musculoskeletal and connective tissue disorders) | 6/54 — Maintenance phase
chest pain (muscular) (Musculoskeletal and connective tissue disorders) | 4/54 — Maintenance phase
pain in legs (Musculoskeletal and connective tissue disorders) | 5/54 — Maintenance phase
hip pain (Musculoskeletal and connective tissue disorders) | 10/54 — Maintenance phase
back pain (Musculoskeletal and connective tissue disorders) | 8/54 — Maintenance phase
arthralgias (Musculoskeletal and connective tissue disorders) | 11/54 — Maintenance phase
neck pain (Musculoskeletal and connective tissue disorders) | 3/54 — Maintenance phase
pain in foot (Musculoskeletal and connective tissue disorders) | 3/54 — Maintenance phase
lower extremity pain (Musculoskeletal and connective tissue disorders) | 6/54 — Maintenance phase
upper extremity pain (Musculoskeletal and connective tissue disorders) | 6/54 — Maintenance phase
knee pain (Musculoskeletal and connective tissue disorders) | 3/54 — Maintenance phase
rash (Skin and subcutaneous tissue disorders) | 10/54 — Maintenance phase
skin darknening (Skin and subcutaneous tissue disorders) | 5/54 — Maintenance phase
pruritus (Skin and subcutaneous tissue disorders) | 4/54 — Maintenance phase
dry skin (Skin and subcutaneous tissue disorders) | 7/54 — Maintenance phase
blurry vision (Eye disorders) | 5/54 — Maintenance phase
bradycardia (Cardiac disorders) | 5/54 — Maintenance phase
genitourinary frequency (Renal and urinary disorders) | 3/54 — Maintenance phase
lung infection (Respiratory, thoracic and mediastinal disorders) | 3/54 — Maintenance phase
cough (Respiratory, thoracic and mediastinal disorders) | 13/54 — Maintenance phase
sore throat (Respiratory, thoracic and mediastinal disorders) | 3/54 — Maintenance phase
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9/54 — Maintenance phase
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7/54 — Maintenance phase
URI (Infections and infestations) | 22/54 — Maintenance phase
skin Infection (Infections and infestations) | 4/54 — Maintenance phase
ear infection (Infections and infestations) | 3/54 — Maintenance phase
fall (Injury, poisoning and procedural complications) | 4/54 — Maintenance phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No